CLINICAL TRIAL: NCT06149624
Title: Supervised Treadmill Intervention to Reduce Inflammation and Depression Through Exercise in HIV: The STRIDE Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MED-2023-32453
Record Dates: First submitted 2023-10-29; First posted 2023-11-29 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Depression; Hiv
MeSH Terms: conditions — Depression; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Placebo Comparator): participants randomized to control group
  Interventions: Behavioral: upfront advice to walk
- Intervention group (Experimental): participants randomized to intervention group
  Interventions: Behavioral: Supervised exercise

INTERVENTIONS:
Behavioral: upfront advice to walk — Control participants will be given upfront advice to walk and also given the wearable activity monitor (Fitbit) and asked to record the total steps achieved each day in a provided log book.
  Arms: control
Behavioral: Supervised exercise — The onsite physiotherapist will also be trained in appropriate supervision and monitoring of exercise therapy in participants with HIV. This training will include titration of the exercise prescription to ensure safe progress is achieved. Participants will be scheduled to come to Mildmay 2 times per week for eight weeks to perform treadmill walking exercise. Intensity will be regulated using 40-60% of heart rate reserve. Additionally, ratings of perceived exertion via the Adult OMNI Walk/Run Scale will be used to guide the intensity of exercise subjectively at a moderate level. The exercise dose participants complete are standard prescriptions for participants with HIV, according to the American College of Sports Medicine.19 The physiotherapist will document the total steps achieved, including the supervised treadmill sessions and activity completed outside the supervised exercise setting (provided by participants via a log book).
  Arms: Intervention group

SUMMARY:
Depression in people living with HIV is associated with worse care engagement, drug adherence, and higher rates of pre-mature mortality. The prevalence of depression is three times greater in those with HIV than comparable controls. While antiretroviral therapy (ART) enables immune reconstitution, those with depression do worse clinically than those without depression even when controlling for HIV stage. However, treating depression in HIV-infected persons is challenging. Even among those virologically suppressed on ART, a significant percentage are resistant to standard pharmacotherapy or psychotherapy for depression. The reasons for this are complex and poorly understood. An emerging body of evidence indicates that inflammation may perpetuate depression. Given people with HIV have ongoing increased inflammation, this could help explain part of why depression rates are so high in people with HIV.

Treatments for HIV-associated depression would likely be more effective if they were anti- inflammatory in nature. One possible treatment is exercise. Exercise is acutely pro-inflammatory due to catabolism but in the long term is anti-inflammatory. However, few studies have investigated exercise as a treatment for HIV-associated depression. The study objective is to perform a feasibility study to evaluate a larger trial evaluating the efficacy of exercise as an intervention for depression in people with HIV.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Mildmay HIV clinic
* Adults 18-45 years old
* HIV positive
* Receiving HIV therapy
* HIV viral suppression (<400 copies/mL) per chart review
* Mild to Moderate (PHQ9 score >5 but >20)
* Not currently engaged in a formal exercise program or manual labor such as construction or delivery requiring a manual bike or walking
* Able to walk/run on a treadmill
* Informed consent

Exclusion Criteria:

* Women pregnant or breastfeeding
* Suicidal (PHQ-9 question 9 score >2) or Severely Depressed (PHQ-9 score >20)
* Uncontrolled hypertension (≥180 systolic or ≥100 diastolic blood pressure)
* Lower limb orthopedic limitations (e.g. amputations, arthritis)
* Resting heart rate >90/min
* Known atherosclerotic or non-atherosclerotic peripheral artery disease.
* Exercise intolerance due to other known medical condition(s) which may make it unsafe for the patients to participate in.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Percent completion of the prescribed aerobic exercise intervention | 8 weeks
  assessed by research staff logging participation

SECONDARY OUTCOMES:
acceptability of the intervention | 8 weeks
  assessed via post intervention survey
feasibility of using a wearable exercise tracker 2 | 8 weeks
  calories burned during the intervention period among Ugandans with HIV and depression
feasibility of using a wearable exercise tracker 1 | 8 weeks
  assess the volume of exercise based on steps achieved, during the intervention period among Ugandans with HIV and depression
effect size | baseline and 8 weeks
  - measure the mean and standard deviation of baseline and 8-week serum BDNF level to estimate an effect size
effect size | baseline and 8 weeks
  - measure the mean and standard deviation of baseline and 8-week serum IL-6 level to estimate an effect size
power estimate | baseline and 8 weeks
  - measure the mean and standard deviation of baseline and 8-week serum BDNF to power a future study
power estimate | baseline and 8 weeks
  - measure the mean and standard deviation of baseline and 8-week serum IL-6 level to power a future study
depression score | baseline and 8 weeks
  depression score via PHQ-9
aerobic fitness | Baseline and 8 weeks
  measure the mean aerobic fitness at baseline and at 8 weeks measured via METS/watts achieved
aerobic fitness | Baseline and 8 weeks
  measure the total time/distance achieved
effect size for a future intervention | Baseline and 8 weeks
  measure the mean and standard deviation for total time/distance to estimate the effect size for a future intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Lofgren, PhD, Principal Investigator — University of Minnesota; Ryan Mays, PhD, Principal Investigator — University of Minnesota; Anita Arinda, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States